CLINICAL TRIAL: NCT02193373
Title: What is the Best Osteopathic Manipulative Medicine (OMM) Approach to Affect Autonomic Nervous System (ANS) Control of Heart Rate Variability (HRV)?
Brief Title: Study of Osteopathic Manipulative Medicine on the Autonomic Nervous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: BHS-1044
Record Dates: First submitted 2014-07-15; First posted 2014-07-17 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Osteopathic Manual Manipulation of Neurovascular Regulation
Keywords: Osteopathic Manipulative Medicine; Autonomic Nervous System; Heart Rate Variability; Sub-Occipital Release; Rib-Raising; Stellate Ganglion Release
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Sub-Occipital Release (Active Comparator): Osteopathic Manual Medicine
  Interventions: Other: Osteopathic Manual Medicine
- Rib-Raising (Active Comparator): Osteopathic Manual Medicine
  Interventions: Other: Osteopathic Manual Medicine
- Stellate Ganglion Release (Active Comparator): Osteopathic Manual Medicine
  Interventions: Other: Osteopathic Manual Medicine
- All techniques (Active Comparator): Osteopathic Manual Medicine
  Interventions: Other: Osteopathic Manual Medicine
- All Techniques-S (Sham Comparator): Sham Osteopathic Manual Medicine
  Interventions: Other: Sham
- Sub-Occipital Release-S (Sham Comparator): Sham Osteopathic Manual Medicine
  Interventions: Other: Sham
- Rib-Raising-S (Sham Comparator): Sham Osteopathic Manual Medicine
  Interventions: Other: Sham
- Stellate Ganglion Release -S (Sham Comparator): Sham Osteopathic Manual Medicine
  Interventions: Other: Sham

INTERVENTIONS:
Other: Osteopathic Manual Medicine — Osteopathic Manual Medicine
  Other Names: Sub-Occipital Release; Rib-Raising; Stellate Ganglion Release
  Arms: All techniques; Rib-Raising; Stellate Ganglion Release; Sub-Occipital Release
Other: Sham — Osteopathic Manual Medicine
  Other Names: Sham sub-occipital release; Sham stellate ganglion release; Sham rib raising
  Arms: All Techniques-S; Rib-Raising-S; Stellate Ganglion Release -S; Sub-Occipital Release-S

SUMMARY:
The purpose this study is to determine which manual medicine technique or combination of techniques has the greatest effect on the natural changes in heart rate.

DETAILED DESCRIPTION:
This study intends to examine how three different OMM techniques, sub-occipital release, rib-raising, and stellate ganglion release, impact autonomic nervous system tone. Subjects will be randomly assigned to one of four cohort groups, receiving either sub-occipital release, rib-raising, stellate ganglion release or all three treatment techniques. A shift towards sympathetic tone will be induced in all subjects using a tilted-to-seated-position test (Tilt-Seated Position test) and cognitive challenge test, consisting of computerized questions that become progressively more difficult, and which subjects are asked to answer as quickly and accurately as possible. These stress tests will be induced twice, once without any OMM treatment and a second time with the designated OMM treatment(s). The sympathetic-dependent response to orthostatic change and cognitive challenges will be determined by Fourier analysis of heart rate variability, recorded using an EKG attached to each subject.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Individual capable of giving consent between the ages of 20-50
* Normal blood pressure as defined by the Seventh Report of US National Committee on Prevention, Detection, Education and Treatment of High Blood Pressure
* Normal EKG
* Normal Heart Rate

Exclusion Criteria:

* Chronic Cardiovascular Disease (including but not limited to: congestive heart failure, previous myocardial infarction, any cardiomyopathy, any arrhythmia, or previous cardiac surgery)
* Hypertension as defined by the Seventh Report of US National Committee on Prevention, Detection, Education and Treatment of High Blood Pressure or hypertensive medications
* Smoking
* Asthma
* Pregnancy
* Diabetes
* Current or recent illness (within the past 7 days)
* Any manipulative therapies within the previous 7 days (including but not limited to: osteopathic manipulative treatment, massage or acupuncture)
* Well conditioned athletes (such as long distance runners)
* Anyone who fails to have an increased heart rate with the passive tilt test (50 degrees head-up)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2014-06; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change in Heart Rate Variability | one hour
  The participant will lay on a table with electrocardiogram leads recording heart rate while an investigator manually engages the soft tissue on different areas of the participant's head, neck, or back.

SECONDARY OUTCOMES:
Effect of Diet and sleep on Heart Rate Variability | Three days
  heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Jayme D Mancini, PhD, DO, Principal Investigator — New York Institute of Technology, College of Osteopathic Medicine; Theodore Flaum, DO, Principal Investigator — New York Institute of Technology, College of Osteopathic Medicine
Locations (1):
- New York Institute of Technology College of Osteopathic Medicine Academic Health Care Center, Old Westbury, New York, United States

REFERENCES:
- [Background] Henderson AT, Fisher JF, Blair J, Shea C, Li TS, Bridges KG. Effects of rib raising on the autonomic nervous system: a pilot study using noninvasive biomarkers. J Am Osteopath Assoc. 2010 Jun;110(6):324-30. PMID 20606239
- [Background] Shi X, Rehrer S, Prajapati P, Stoll ST, Gamber RG, Downey HF. Effect of cranial osteopathic manipulative medicine on cerebral tissue oxygenation. J Am Osteopath Assoc. 2011 Dec;111(12):660-6. PMID 22182951